CLINICAL TRIAL: NCT06367933
Title: Mini-invasive Fusion in Spine Surgery for Neuromuscolar Scoliosis: a Pilot Study
Brief Title: Mini-invasive Spine Surgery for Neuromuscolar Scoliosis
Acronym: MISNM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISNM
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Neuromuscular Scoliosis; Spine Deformity; Surgery; Vertebral Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): severe neuromuscolar scoliosis who need surgical correction
  Interventions: Procedure: mini-invasive spine surgery

INTERVENTIONS:
Procedure: mini-invasive spine surgery — spine deformity correction using a mini-invasive technique

SUMMARY:
Neuromuscular scoliosis (SNM) are deformities related to the impairment of normal function of the central nervous system (CNS) and/or peripheral nervous system (PNS) resulting in alterations to the of the functional unit represented by the integrated motor sequence (SIM). At the level of the spine, dysfunction of the SIM results in altered dynamic support of the spine. This results in a control of the trunk that is not harmonious due to the lack of effective mechanisms of muscle compensation. In particular, a greater degree of pelvic tilt with respect to the ground plane, with an increase in the degree of the so-called pelvic obliquity (OP), a fundamental parameter in walking and maintaining the seated posture. Spinal deformity causes severe alterations of the rib cage resulting in respiratory failure that often requires ventilatory supports and is associated with frequent airway infections, including pneumonias, often fatal. SNMs also express other comorbidities: cardiac (heart failure), neurological (epilepsy), nutritional that necessitate careful management multidisciplinary and especially anesthesiological evaluation for the peri-operative management. The surgical treatment of SNM constitutes a topic that is still debated due to both the bio-mechanical peculiarities of SNM and the clinical features, particularly comorbidities, that characterize this patient population. Compared with idiopathic scoliosis surgery, in SNM there is a higher rate of complications. To date, most of the complications are respiratory in nature (23%), followed by complications mechanical of the implanted surgical instrumentation (13%), and surgical site infections (11%). Furthermore, there is evidence that SNM surgery correlates with increased blood loss intraoperative. To date, it is recognized in the literature that the safest and most effective surgical treatment for SNMs is arthrodesis posterior instrumented with pedicle screws extended to the pelvis. In the years, mini-invasive surgical techniques have become increasingly prominent. invasive with the goal of reducing operative time, blood loss and complications themselves.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SNM
* Age 9 to 25 years
* Male and female gender
* Preoperative Cobb > 45° COBB
* Preoperative pelvic obliquity > 10°
* Extent of scoliotic curve (expressed in COBB degrees) on supine whole spine X-ray

  ≤ 25% compared with magnitude of curve assessed on into spinal X-rays from supine sitting.
* Loss of walking ability
* Absence of emergency criteria for spinal surgery

Exclusion Criteria:

* Scoliosis with etiology other than SNM
* Pre-operative Cobb < 45° COBB
* Preoperative pelvic obliquity < 10°
* High anesthesiologic risk for severe respiratory deficit
* Criteria for surgical urgency
* Preserved ambulatory capacity
* Patients who did not perform follow-up at the Rizzoli Orthopaedic Institute;
* Patients whose parents/guardians have denied consent for access to their own medical records.
* Language barrier

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | At baseline (Day 0)
  The VAS scale is an objective method of pain measurement
Visual Analogue Scale | At 12 month follow-up
  The VAS scale is an objective method of pain measurement
Spine Correction | 12 months
  The correction of the curvature of the back will be evaluated via x-ray
Spine Correction | 24 months
  The correction of the curvature of the back will be evaluated via x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Modi HN, Hong JY, Mehta SS, Srinivasalu S, Suh SW, Yi JW, Yang JH, Song HR. Surgical correction and fusion using posterior-only pedicle screw construct for neuropathic scoliosis in patients with cerebral palsy: a three-year follow-up study. Spine (Phila Pa 1976). 2009 May 15;34(11):1167-75. doi: 10.1097/BRS.0b013e31819c38b7. PMID 19444065